CLINICAL TRIAL: NCT00768781
Title: Augmenting Behavior Therapy for Insomnia With Mindfulness Meditation
Brief Title: Mindfulness-Based Approaches to Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Stanford University (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Jason C. Ong, PhD, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23AT003678 (NIH); K23AT003678 (NIH)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Insomnia
Keywords: insomnia; hyperarousal; mindfulness meditation; complementary and alternative medicine; cognitive-behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mindfulness-Based Stress Reduction; Waiting Lists; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness-Based Stress Reduction (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Mindfulness-Based Therapy for Insomnia (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Therapy for Insomnia
- Behavioral Therapy for Insomnia (Delayed treatment condition) (Other)
  Interventions: Behavioral: Wait-List + Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The rationale for treatment is that MBSR targets arousal, which is a prominent perpetuating factor of insomnia. Each session meets weekly for 120 minutes and consists of a therapist-led mindfulness meditation, followed by a discussion of the meditation and its application into the participant's everyday life. For homework, each participant is required to practice formal meditation at least 45 minutes a day, 6 days per week. Participants will be provided a tape, an mp3 file, or CD to aid in the participant's personal practice at home. Formal meditations that will be led and discussed include eating meditation, body scan, sitting meditation, Hatha Yoga, and walking meditation. In addition, informal mindfulness practices will be discussed.
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Mindfulness-Based Therapy for Insomnia — MBTI treatment includes the hypothesized active elements of both mindfulness meditation and behavior therapy for insomnia. The intervention includes 8 weekly sessions. Each session meets weekly for approximately 120 minutes. The general format of each session includes formal mindfulness meditation (quiet and movement meditations) and instructions for the behavioral intervention, with a focus on integrating the principles of mindfulness with these instructions. Each participant is required to practice formal meditation for at least 45 minutes a day, 6 days per week as homework. Participants are provided a tape, mp3 file, or CD to aid in the participant's personal practice at home.
  Arms: Mindfulness-Based Therapy for Insomnia
Behavioral: Wait-List + Behavioral Therapy for Insomnia — This delayed treatment condition consists of an 8-week monitoring period (sleep diaries, PSAS) and then BT. The BT treatment consists of 8 sessions of behavioral interventions for insomnia, with instructions targeting the nighttime symptoms of insomnia. The primary components of this treatment package are stimulus control, sleep restriction, and sleep hygiene education. In the BT condition, each weekly session lasts 120 minutes and consists of formal instructions for the behavioral interventions along with a time for discussion of the application of these instructions into each participant's unique circumstances.
  Arms: Behavioral Therapy for Insomnia (Delayed treatment condition)

SUMMARY:
The overall goal of this project is to evaluate the evidence for the efficacy of two mindfulness-based interventions, mindfulness-based therapy for insomnia (MBT-I) and mindfulness-based stress reduction (MBSR), for reducing arousal and improving sleep among individuals with psychophysiological insomnia.

Specific Aim 1: To obtain evidence for the relative effects of MBT-I and MBSR compared to a delayed-treatment control condition followed by behavior therapy for insomnia (BT-I) on arousal levels. It is hypothesized that MBSR and MBT-I will be superior to the control condition at reducing arousal levels.

Specific Aim 2: To obtain evidence for the relative effects of MBT-I, MBSR, and the delayed-treatment control on sleep. It is hypothesized that MBT-I will be superior to the MBSR and control conditions at improving sleep parameters.

Specific Aim 3: To investigate the relationship between measures of arousal (self-report and objective measures) and sleep (self-report and objective measures) to enhance the understanding of the role of arousal in psychophysiological insomnia.

DETAILED DESCRIPTION:
The conceptual model for this study identifies two possible targets of treatment: arousal and sleep. In this model, BT for insomnia directly targets nighttime symptoms of insomnia (BT pathway), which improves sleep by increasing the homeostatic drive for sleep. Although BT is hypothesized to indirectly reduce arousal, no study has specifically investigated this effect. In contrast, MBSR is an intervention that is hypothesized to target arousal and, as preliminary findings suggest, also improves some symptoms of insomnia (MBSR pathway). It is therefore hypothesized that a combination of BT and mindfulness is superior to each treatment alone as it targets both nighttime symptoms and hyperarousal (Mindfulness + BT pathway). Our preliminary data suggests that this combination treatment has effects on both self-reported arousal and sleep. Conceptually, this novel approach would provide a set of self-regulating skills that could potentially target a broader range of daytime and nighttime symptoms that is characteristic of an insomnia disorder.

To test the conceptual model, this study employs a randomized clinical trial design with three conditions: 1) Mindfulness-Based Therapy for insomnia (MBT-I), 2) mindfulness-based stress reduction (MBSR), and 3) delayed-treatment condition followed by behavior therapy for insomnia (BT-I). Each of the three treatments will be delivered in a group format with 8 weekly sessions spanning an 8-week period.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for psychophysiological insomnia
* Males and females of age 21 or older

Exclusion Criteria:

* Unstable medical condition that is known to impact sleep
* Psychiatric conditions likely to impact the practice of meditation
* Current active suicidal ideation
* Presence of a primary sleep disorder other than primary insomnia
* Evidence of paradoxical insomnia
* Evidence of idiopathic insomnia
* Frequent use of alcohol at bedtime
* Excessive daily caffeine consumption
* Current use of sleep medications on a regular basis
* Inadequate proficiency in English
* Inability to commit to attending therapy sessions due to schedule conflicts
* Women who are pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pre-Sleep Arousal Scale (PSAS) total score | Baseline, during txt, post-txt, 3 month follow-up, 6 month follow-up
Sleep Diaries (Total Wake Time) | Baseline, post-txt, 6 month follow-up

SECONDARY OUTCOMES:
Actigraphy measures of sleep/wake time | Baseline, during txt, post-txt, 3 month follow-up, 6 month follow-up
Polysomnographic measures of sleep parameters | Baseline, post-txt, 6 month follow-up
Insomnia Severity Index (ISI) total score | Baseline, post-txt, 3 month follow-up, 6 month follow-up
Five Factor Questionnaire (Mindfulness Skills) Total score | Baseline, post-txt, 3 month follow-up, 6 month follow-up
Dysfunctional Beliefs and Attitudes about Sleep (DBAS) score | Baseline, post-txt, 3 month follow-up, 6 month follow-up
Hyperarousal Scale (HAS) score | Baseline, post-txt, 3 month follow-up, 6 month follow-up
Heart Rate variability (HR) | Baseline, post-treatment, 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jason C Ong, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Sleep Disorders Center, Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Goldstein MR, Turner AD, Dawson SC, Segal ZV, Shapiro SL, Wyatt JK, Manber R, Sholtes D, Ong JC. Increased high-frequency NREM EEG power associated with mindfulness-based interventions for chronic insomnia: Preliminary findings from spectral analysis. J Psychosom Res. 2019 May;120:12-19. doi: 10.1016/j.jpsychores.2019.02.012. Epub 2019 Feb 28. PMID 30929703
- [Derived] Ong JC, Manber R, Segal Z, Xia Y, Shapiro S, Wyatt JK. A randomized controlled trial of mindfulness meditation for chronic insomnia. Sleep. 2014 Sep 1;37(9):1553-63. doi: 10.5665/sleep.4010. PMID 25142566